CLINICAL TRIAL: NCT06237699
Title: Diary Implementation as a Prelude to Integrated Interventions in Person-centered Care in the Intensive Care Unit
Brief Title: Effects of a Digital Diary on the Psychological Well-being of Former ICU Patients.
Acronym: DIPIC
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Erwin Ista, Associate professor, Erasmus Medical Center
Other Study IDs: MEC-2022-0580
Record Dates: First submitted 2024-01-06; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Depression, Anxiety; Post Traumatic Stress Disorder; Quality of Life
Keywords: Quality of care; Digital ICU Diary; ICU survivors; Relatives
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ICU survivors without an ICU diary
- ICU relatives without an ICU diary
- ICU survivors with a digital ICU diary
  Interventions: Other: Digital ICU diary
- ICU relatives with a digital ICU diary
  Interventions: Other: Digital ICU diary

INTERVENTIONS:
Other: Digital ICU diary — A digital ICU diary is an electronic platform or application designed to facilitate the documentation and communication of the experiences, progress, and medical journey of patients in the Intensive Care Unit (ICU).
  Groups: ICU relatives with a digital ICU diary; ICU survivors with a digital ICU diary

SUMMARY:
Previous research on the impact of a diary on mental symptoms of PICS, PICS-F, and quality of life in former ICU patients and their relatives has focused specifically on a paper diary. While there has been research on the experiences of former ICU patients, relatives, and ICU nurses regarding the use of a digital diary, it is not known whether this diary has an impact on the psychological well-being and quality of life of former ICU patients and their relatives. A successful implementation of [the digital diary] enables this research. The aim of this study is, therefore, to provide an initial impression of the health-related effects of a digital diary on former ICU patients and their relatives.

DETAILED DESCRIPTION:
Objective: Exploring health-related effects of a digital ICU diary in former ICU patients and their relatives.

Research question 1: What is the effect of a digital ICU diary on the psychological well-being and quality of life in former ICU patients and their relatives? Research question 2: What is the effect of a digital ICU diary on the perceived quality of care and satisfaction with the ICU admission among relatives of former ICU patients?

ELIGIBILITY:
Inclusion criteria for former ICU patients and their relatives:

* Capacity to make decisions autonomously
* Proficiency in the Dutch language
* 18 years of age or older
* ICU length of stay >48 hours
* No use of an ICU diary before (pre-measurement)
* Used the digital Post-IC diary for more than 1 day (post-measurement)

Exclusion criteria for former ICU patients and their relatives:

* Insufficient proficiency in the Dutch language to express themselves on the subject.
* Patients with a pre-admission diagnosis of psychosis or dementia.
* Use of a paper ICU diary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former ICU patients (ICU survivors) & Relatives of (former) ICU patients
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Post Traumatic Stress Disorder (PTSD) [IES-R] | 1-3 months after ICU admission
  PTSD-related symptoms measured with the IMPACT OF EVENTS SCALE-Revised (IES-R)
Number of participants with Anxiety or Depression-related symptoms [HADS] | 1-3 months after ICU admission
  Anxiety-related and depression-related symptoms measured with Hospital Anxiety and Depression Scale (HADS)
The participants' level of quality of life [SF36] | 1-3 months after ICU admission
  The participants' level of quality of life measured with 36-Item Short Form Health Survey SF-36

SECONDARY OUTCOMES:
Relatives' perspectives on the quality of care [CQI-R] | 1 month after ICU admission
  Relatives' perspectives on quality of care and satisfaction measured with Consumer Quality Index- Relatives (CQI-R)

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Erasmus University medical center, Rotterdam, South Holland
  - Medisch Spectrum Twente, Enschede
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Elisabeth-TweeSteden ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided
We ask the participants permission if other studies can you the data also